CLINICAL TRIAL: NCT07243106
Title: Role of Airway Ultrasonography in Predicting Difficult Airway: Comparison of Clinical and Sonographic Parameters
Brief Title: Airway Ultrasound vs Clinical Predictors for Difficult Airway
Status: Not yet recruiting | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 25-MOBAEK-329
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Ultrasonography; Difficult Airway; Preoperative Evaluation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients scheduled for elective surgery under general anesthesia with endotracheal intubation: Demographic data of all participants-including age, sex, type of planned surgery, ASA physical status, and comorbidities-will be recorded. Before induction of anesthesia, all patients will be evaluated using standard clinical airway assessment parameters. These include the Mallampati score, thyromental distance, sternomental distance, neck circumference, and upper lip bite test. Body mass index (BMI) and waist-to-hip ratio will also be measured and documented.
  In the preoperative period, all patients will undergo airway ultrasonography performed by an anesthesiologist. Sonographic assessments will be carried out by a single experienced anesthesiologist using a linear transducer, with the patient positioned in the sniffing position. The following ultrasound measurements will be obtained and recorded: Skin-to-epiglottis distance, skin-to-hyoid bone distance, skin-to-anterior commissure of the vocal cords distance, skin-to-trachea distance at the suprasternal notch level.

SUMMARY:
This prospective observational study aims to evaluate the diagnostic value of airway ultrasonography in predicting difficult intubation in adult patients undergoing elective surgery under general anesthesia. Preoperative sonographic measurements of upper airway structures will be compared with conventional clinical airway assessment parameters such as the Mallampati score, thyromental distance, and sternomental distance.

The study seeks to determine whether ultrasonographic measurements can serve as independent predictors of difficult airway and whether combining them with clinical parameters improves diagnostic accuracy. Additionally, the correlation between sonographic findings and the Intubation Difficulty Scale (IDS) will be analyzed to assess the potential clinical utility of airway ultrasound in preoperative airway evaluation.

DETAILED DESCRIPTION:
Airway management is one of the most critical and potentially life-threatening procedures in anesthesiology practice. Difficult intubation may result in severe morbidity and mortality if not promptly and effectively managed. Therefore, reliable preoperative prediction of a difficult airway is crucial for ensuring patient safety and optimizing perioperative outcomes.

Traditional clinical assessment methods-such as the Mallampati classification, thyromental distance, and sternomental distance-are commonly used to predict difficult airway. However, these predictors have limited sensitivity and specificity, and their diagnostic accuracy may vary depending on operator experience and subjective interpretation.

In recent years, ultrasonography has gained increasing acceptance in anesthesiology as a non-invasive, rapid, inexpensive, and real-time imaging technique. Airway ultrasonography enables direct visualization of individual anatomical variations in the upper airway, providing more objective and reproducible data for airway assessment.

The primary objective of this study is to determine the diagnostic performance of ultrasonographic parameters obtained from preoperative airway ultrasound in predicting difficult laryngoscopy and intubation, and to compare them with conventional clinical assessment methods. The study will also evaluate whether ultrasonographic measurements are independent predictors of difficult airway and whether combining sonographic and clinical parameters enhances overall diagnostic accuracy.

Furthermore, the relationship between ultrasound-based anatomical measurements and the Intubation Difficulty Scale (IDS) will be analyzed. This correlation aims to demonstrate the potential contribution of airway ultrasonography to clinical decision-making and its possible role in improving airway safety in anesthetic practice.

Hypotheses:

H0 (Null Hypothesis): Airway ultrasonography does not provide higher diagnostic accuracy than traditional clinical assessment methods in predicting difficult intubation and has no significant correlation with the Intubation Difficulty Scale (IDS).

H1 (Alternative Hypothesis): Airway ultrasonography provides higher diagnostic accuracy than traditional clinical assessment methods in predicting difficult intubation and is significantly correlated with the Intubation Difficulty Scale (IDS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-60 years
* Scheduled for elective surgery
* ASA (American Society of Anesthesiologists) physical status I, II, or III
* Planned for endotracheal intubation under general anesthesia

Exclusion Criteria:

* Patients requiring emergency surgery
* Patients with a known history of difficult intubation
* Patients with head or neck trauma
* Patients with a history of previous head or neck surgery or head/neck malignancy
* Pregnant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult patients aged 18-60 years, classified as ASA I-III, scheduled for elective surgery under general anesthesia with planned endotracheal intubation. Both male and female patients meeting inclusion criteria and without any exclusion criteria (emergency surgery, known difficult intubation, head/neck trauma, prior head/neck surgery or malignancy, pregnancy) will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The Intubation Difficulty Scale (IDS) | During tracheal intubation (approximately 1-3 minutes after induction of anesthesia)
  The Intubation Difficulty Scale (IDS) is a quantitative scoring system used to objectively assess the complexity of tracheal intubation. It incorporates seven parameters: number of intubation attempts, number of operators, number of alternative techniques used, Cormack-Lehane grade, lifting force required, necessity of external laryngeal pressure, and position of the vocal cords.
  The total IDS score is calculated as the sum of these variables, providing a numerical indicator of intubation difficulty (IDS = 0 indicates easy intubation; IDS = 1-5 mild to moderate difficulty; IDS > 5 difficult intubation).
Difficulty of mask ventilation | During 2-minute face mask ventilation after induction of anesthesia
  After standard induction of anesthesia, all patients will be ventilated via face mask for 2 minutes, followed by tracheal intubation using a Macintosh laryngoscope. The difficulty of mask ventilation will be assessed using the Han Mask Ventilation Scale, defined as follows:
  Class 1: Mask ventilation possible
  Class 2: Mask ventilation possible with the use of an oral airway or other adjuncts
  Class 3: Mask ventilation possible only with the assistance of a second person
  Class 4: Mask ventilation impossible

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared with other researchers upon reasonable request
Supporting Information: Study Protocol, SAP